CLINICAL TRIAL: NCT02455726
Title: Magnesium Oral Supplementation to Reduce Pain in Patients With Severe Peripheral Arterial Occlusive Disease: The MAG-PAPER Randomized Clinical Trial
Brief Title: Magnesium Oral Supplementation to Reduce Pain Inpatients With Severe Peripheral Arterial Occlusive Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Monica Aida Venturini, MD, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1601 gluta-aos
Record Dates: First submitted 2015-04-23; First posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Magnesium Oxide; Pain
MeSH Terms: conditions — Peripheral Arterial Disease; Pain | interventions — Magnesium Oxide; Fructose; Oxycodone; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mg-group (Experimental): Standard therapy plus magnesium oxide.
  * Standard therapy: oxycodone 5 mg and pregabalin 25 mg per day for two weeks. Starting by day 2, the opioid dose will be titrated every 48 hours in order to reach the maximum therapeutic goal and to minimize side effects.
  * A rescue dose: paracetamol 1g (maximum dose 3 g per day).
  Interventions: Dietary Supplement: Magnesium oxide; Drug: Oxycodone; Drug: Pregabalin
- C-group (Placebo Comparator): Standard therapy plus fructose.
  * Standard therapy: oxycodone 5 mg and pregabalin 25 mg per day for two weeks. Starting by day 2, the opioid dose will be titrated every 48 hours in order to reach the maximum therapeutic goal and to minimize side effects.
  * A rescue dose: paracetamol 1g (maximum dose 3 g per day).
  Interventions: Dietary Supplement: Fructose; Drug: Oxycodone; Drug: Pregabalin

INTERVENTIONS:
Dietary Supplement: Magnesium oxide — Oral magnesium oxide 300 mg twice a day
  Arms: Mg-group
Dietary Supplement: Fructose — Oral fructose 10 g twice a day
  Arms: C-group
Drug: Oxycodone — Oxycodone hydrochloride 5 mg at 8 am
  Other Names: Oxycontin, Mundipharma Pharmaceutic
Drug: Pregabalin — Pregabalin 25 mg at 8 pm
  Other Names: Lyrica, Pfizer Italia

SUMMARY:
Magnesium exerts analgesic effects in several animal pain models and in patients affected by acute postoperative pain and chronic pain of neuropathic origin. There is no evidence that magnesium can modulate pain in patients with peripheral arterial occlusive disease (PAOD).

We describe the protocol of a single-center randomized double-blind clinical trial aimed at assessing the efficacy of oral magnesium supplementation in controlling severe pain in patients with advanced PAOD.

DETAILED DESCRIPTION:
* Adult patients admitted to our Acute Pain Service for intractable pain will be eligible if they are affected by PAOD at stages III and IV of Lèriche-Fontaine classification, and are opioid-naïve.
* Patients enrolled will be randomized to the control group, treated with standard therapy, consisting of an oral administration of oxycodone 5 mg and pregabalin 25 mg per day plus placebo (fructose 10 g) twice a day for two weeks, or to the experimental group, treated with magnesium oxide 300 mg twice a day.
* Randomization will be computer-generated, with allocation concealment obtained using opaque, sequentially numbered and sealed envelopes. Trials participants, care providers, data collectors, outcome assessors and data analysts will be blinded to treatment allocation.
* Patients will be evaluated on the day of hospital admission (day 0) and on days 2, 4, 6, 8, 12, and 14 with the following information being collected: daily oxycodone dose received; patient's perceived average and maximum pain using the Numerical Rating Scale (NRS: 0=no pain to 10=worst possible pain); pain relief using Pain Relief Scale (PRS: 0% no pain relief to 100% complete pain relief); characteristics of the pain, using the Neuropathic Pain Scale (NPS: 10 items); impact of pain on the patient's daily activities, using the Brief Pain Inventory (BPI; 9 items).
* A sample size calculation performed for the primary outcome showed that 150 patients (75 per group) are needed to achieve 90% power to detect a minimum reduction of 30% in oxycodone dosage in the experimental group, after allowing for a drop-out rate of around 20%.
* Ethical approval of the study protocol has been obtained from Comitato Etico Provinciale di Brescia, Brescia, Italy.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (18 years or above)
* PAOD at stages III and IV according to the Lèriche-Fontaine classification
* no treatment with opioids at the time of recruitment

Exclusion Criteria:

* renal failure (serum creatinine ≥ 2.0 mg/dl);
* congestive heart failure (New York Heart Association, NYHA > 3);
* treatment with digoxin and/or calcium channel blockers;
* pre-existing neuromuscular diseases;
* chronic diarrhea;
* acute limb ischemia successfully treated with interventional angiography, Fogarty embolectomy and/or surgical revascularization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The oxycodone dosage needed to achieve satisfactory analgesia | 14 days
  Patient's satisfactory analgesia is defined as NRS ≤4

SECONDARY OUTCOMES:
Level of pain relief | 2 days
  The level of pain relief is measured using Pain Relief Scale
Time to satisfactory analgesia | from 2 to 14 days
  The time needed to achieve satisfactory analgesia (NRS≤4)
Time to 50% reduction of pain | from 2 to 14 days
  The time needed to achieve a reduction of pain of 50% using Pain Relief Scale(PRS = 50%)

CONTACTS AND LOCATIONS:
Overall Officials: Monica A Venturini, Doctor, Principal Investigator

REFERENCES:
- [Background] Dowell D, Kunins HV, Farley TA. Opioid analgesics--risky drugs, not risky patients. JAMA. 2013 Jun 5;309(21):2219-20. doi: 10.1001/jama.2013.5794. No abstract available. PMID 23700072
- [Background] Fowkes FG, Rudan D, Rudan I, Aboyans V, Denenberg JO, McDermott MM, Norman PE, Sampson UK, Williams LJ, Mensah GA, Criqui MH. Comparison of global estimates of prevalence and risk factors for peripheral artery disease in 2000 and 2010: a systematic review and analysis. Lancet. 2013 Oct 19;382(9901):1329-40. doi: 10.1016/S0140-6736(13)61249-0. Epub 2013 Aug 1. PMID 23915883
- [Background] Iseri LT, French JH. Magnesium: nature's physiologic calcium blocker. Am Heart J. 1984 Jul;108(1):188-93. doi: 10.1016/0002-8703(84)90572-6. No abstract available. PMID 6375330
- [Background] Kew JN, Kemp JA. Ionotropic and metabotropic glutamate receptor structure and pharmacology. Psychopharmacology (Berl). 2005 Apr;179(1):4-29. doi: 10.1007/s00213-005-2200-z. Epub 2005 Feb 25. PMID 15731895
- [Background] Recio-Pinto E, Castillo C. Peripheral N-methyl-D-aspartate receptors as possible targets for chronic pain treatment. Techniques in Reg Anesth & Pain Manag 2010;14:48-58
- [Background] Fisher K, Coderre TJ, Hagen NA. Targeting the N-methyl-D-aspartate receptor for chronic pain management. Preclinical animal studies, recent clinical experience and future research directions. J Pain Symptom Manage. 2000 Nov;20(5):358-73. doi: 10.1016/s0885-3924(00)00213-x. PMID 11068158
- [Background] Hewitt DJ. The use of NMDA-receptor antagonists in the treatment of chronic pain. Clin J Pain. 2000 Jun;16(2 Suppl):S73-9. doi: 10.1097/00002508-200006001-00013. PMID 10870744
- [Background] De Kock MF, Lavand'homme PM. The clinical role of NMDA receptor antagonists for the treatment of postoperative pain. Best Pract Res Clin Anaesthesiol. 2007 Mar;21(1):85-98. doi: 10.1016/j.bpa.2006.12.006. PMID 17489221
- [Background] Petrenko AB, Yamakura T, Baba H, Shimoji K. The role of N-methyl-D-aspartate (NMDA) receptors in pain: a review. Anesth Analg. 2003 Oct;97(4):1108-1116. doi: 10.1213/01.ANE.0000081061.12235.55. PMID 14500166
- [Background] Nechifor M. Magnesium involvement in pain. Magnes Res. 2011 Dec;24(4):220-2. doi: 10.1684/mrh.2011.0296. No abstract available. PMID 22061718
- [Background] Hasanein P, Parviz M, Keshavarz M, Javanmardi K, Mansoori M, Soltani N. Oral magnesium administration prevents thermal hyperalgesia induced by diabetes in rats. Diabetes Res Clin Pract. 2006 Jul;73(1):17-22. doi: 10.1016/j.diabres.2005.12.004. Epub 2006 Jan 18. PMID 16417942
- [Background] Rondon LJ, Privat AM, Daulhac L, Davin N, Mazur A, Fialip J, Eschalier A, Courteix C. Magnesium attenuates chronic hypersensitivity and spinal cord NMDA receptor phosphorylation in a rat model of diabetic neuropathic pain. J Physiol. 2010 Nov 1;588(Pt 21):4205-15. doi: 10.1113/jphysiol.2010.197004. PMID 20837644
- [Background] Begon S, Pickering G, Eschalier A, Dubray C. Magnesium increases morphine analgesic effect in different experimental models of pain. Anesthesiology. 2002 Mar;96(3):627-32. doi: 10.1097/00000542-200203000-00019. PMID 11873038
- [Background] Bujalska M, Makulska-Nowak H, Gumulka SW. Magnesium ions and opioid agonists in vincristine-induced neuropathy. Pharmacol Rep. 2009 Nov-Dec;61(6):1096-104. doi: 10.1016/s1734-1140(09)70172-0. PMID 20081245
- [Background] Ulugol A, Aslantas A, Ipci Y, Tuncer A, Hakan Karadag C, Dokmeci I. Combined systemic administration of morphine and magnesium sulfate attenuates pain-related behavior in mononeuropathic rats. Brain Res. 2002 Jul 5;943(1):101-4. doi: 10.1016/s0006-8993(02)02618-5. PMID 12088843
- [Background] Chen Y, Zhang Y, Zhu YL, Fu PL. Efficacy and safety of an intra-operative intra-articular magnesium/ropivacaine injection for pain control following total knee arthroplasty. J Int Med Res. 2009 Nov-Dec;37(6):1733-41. doi: 10.1177/147323000903700609. PMID 20146871 (Retraction: PMID 23206489 J Int Med Res. 2012;40(5):2031)
- [Background] Bondok RS, Abd El-Hady AM. Intra-articular magnesium is effective for postoperative analgesia in arthroscopic knee surgery. Br J Anaesth. 2006 Sep;97(3):389-92. doi: 10.1093/bja/ael176. Epub 2006 Jul 11. PMID 16835255
- [Background] Cizmeci P, Ozkose Z. Magnesium sulphate as an adjuvant to total intravenous anesthesia in septorhinoplasty: a randomized controlled study. Aesthetic Plast Surg. 2007 Mar-Apr;31(2):167-73. doi: 10.1007/s00266-006-0194-5. PMID 17437152
- [Background] Nechifor M. Magnesium in major depression. Magnes Res. 2009 Sep;22(3):163S-166S. PMID 19780403
- [Background] Murck H. Ketamine, magnesium and major depression--from pharmacology to pathophysiology and back. J Psychiatr Res. 2013 Jul;47(7):955-65. doi: 10.1016/j.jpsychires.2013.02.015. Epub 2013 Mar 26. PMID 23541145
- [Background] Albrecht E, Kirkham KR, Liu SS, Brull R. Peri-operative intravenous administration of magnesium sulphate and postoperative pain: a meta-analysis. Anaesthesia. 2013 Jan;68(1):79-90. doi: 10.1111/j.1365-2044.2012.07335.x. Epub 2012 Nov 1. PMID 23121612
- [Background] Seyhan TO, Tugrul M, Sungur MO, Kayacan S, Telci L, Pembeci K, Akpir K. Effects of three different dose regimens of magnesium on propofol requirements, haemodynamic variables and postoperative pain relief in gynaecological surgery. Br J Anaesth. 2006 Feb;96(2):247-52. doi: 10.1093/bja/aei291. Epub 2005 Nov 25. PMID 16311277
- [Background] Ryu JH, Kang MH, Park KS, Do SH. Effects of magnesium sulphate on intraoperative anaesthetic requirements and postoperative analgesia in gynaecology patients receiving total intravenous anaesthesia. Br J Anaesth. 2008 Mar;100(3):397-403. doi: 10.1093/bja/aem407. PMID 18276652
- [Background] Tramer MR, Schneider J, Marti RA, Rifat K. Role of magnesium sulfate in postoperative analgesia. Anesthesiology. 1996 Feb;84(2):340-7. doi: 10.1097/00000542-199602000-00011. PMID 8602664
- [Background] Song JW, Lee YW, Yoon KB, Park SJ, Shim YH. Magnesium sulfate prevents remifentanil-induced postoperative hyperalgesia in patients undergoing thyroidectomy. Anesth Analg. 2011 Aug;113(2):390-7. doi: 10.1213/ANE.0b013e31821d72bc. Epub 2011 May 19. PMID 21596876
- [Background] Tugrul S, Degirmenci N, Eren SB, Dogan R, Veyseller B, Ozturan O. Analgesic effect of magnesium in post-tonsillectomy patients: a prospective randomised clinical trial. Eur Arch Otorhinolaryngol. 2015 Sep;272(9):2483-7. doi: 10.1007/s00405-014-3219-8. Epub 2014 Aug 6. PMID 25097030
- [Background] Borazan H, Kececioglu A, Okesli S, Otelcioglu S. Oral magnesium lozenge reduces postoperative sore throat: a randomized, prospective, placebo-controlled study. Anesthesiology. 2012 Sep;117(3):512-8. doi: 10.1097/ALN.0b013e3182639d5f. PMID 22797283
- [Background] Brill S, Sedgwick PM, Hamann W, Di Vadi PP. Efficacy of intravenous magnesium in neuropathic pain. Br J Anaesth. 2002 Nov;89(5):711-4. PMID 12393768
- [Background] Crosby V, Wilcock A, Corcoran R. The safety and efficacy of a single dose (500 mg or 1 g) of intravenous magnesium sulfate in neuropathic pain poorly responsive to strong opioid analgesics in patients with cancer. J Pain Symptom Manage. 2000 Jan;19(1):35-9. doi: 10.1016/s0885-3924(99)00135-9. PMID 10687324
- [Background] Suresh S, Lozono S, Hall SC. Large-dose intravenous methotrexate-induced cutaneous toxicity: can oral magnesium oxide reduce pain? Anesth Analg. 2003 May;96(5):1413-1414. doi: 10.1213/01.ANE.0000057140.33744.65. PMID 12707144
- [Background] Kroin JS, McCarthy RJ, Von Roenn N, Schwab B, Tuman KJ, Ivankovich AD. Magnesium sulfate potentiates morphine antinociception at the spinal level. Anesth Analg. 2000 Apr;90(4):913-7. doi: 10.1097/00000539-200004000-00025. PMID 10735798
- [Background] Yousef AA, Al-deeb AE. A double-blinded randomised controlled study of the value of sequential intravenous and oral magnesium therapy in patients with chronic low back pain with a neuropathic component. Anaesthesia. 2013 Mar;68(3):260-6. doi: 10.1111/anae.12107. Epub 2012 Dec 17. PMID 23384256
- [Background] Lysakowski C, Dumont L, Czarnetzki C, Tramer MR. Magnesium as an adjuvant to postoperative analgesia: a systematic review of randomized trials. Anesth Analg. 2007 Jun;104(6):1532-9, table of contents. doi: 10.1213/01.ane.0000261250.59984.cd. PMID 17513654
- [Background] Pickering G, Morel V, Simen E, Cardot JM, Moustafa F, Delage N, Picard P, Eschalier S, Boulliau S, Dubray C. Oral magnesium treatment in patients with neuropathic pain: a randomized clinical trial. Magnes Res. 2011 Jun;24(2):28-35. doi: 10.1684/mrh.2011.0282. PMID 21659058
- [Background] Felsby S, Nielsen J, Arendt-Nielsen L, Jensen TS. NMDA receptor blockade in chronic neuropathic pain: a comparison of ketamine and magnesium chloride. Pain. 1996 Feb;64(2):283-291. doi: 10.1016/0304-3959(95)00113-1. PMID 8740606
- [Background] Mikkelsen S, Dirks J, Fabricius P, Petersen KL, Rowbotham MC, Dahl JB. Effect of intravenous magnesium on pain and secondary hyperalgesia associated with the heat/capsaicin sensitization model in healthy volunteers. Br J Anaesth. 2001 Jun;86(6):871-3. doi: 10.1093/bja/86.6.871. PMID 11573598
- [Background] Ruger LJ, Irnich D, Abahji TN, Crispin A, Hoffmann U, Lang PM. Characteristics of chronic ischemic pain in patients with peripheral arterial disease. Pain. 2008 Sep 30;139(1):201-208. doi: 10.1016/j.pain.2008.03.027. Epub 2008 May 9. PMID 18472216
- [Background] Shechter M, Bairey Merz CN, Stuehlinger HG, Slany J, Pachinger O, Rabinowitz B. Effects of oral magnesium therapy on exercise tolerance, exercise-induced chest pain, and quality of life in patients with coronary artery disease. Am J Cardiol. 2003 Mar 1;91(5):517-21. doi: 10.1016/s0002-9149(02)03297-6. PMID 12615252
- [Background] FONTAINE R, KIENY R, GANGLOFF JM, CUNY A, SUHLER A, GONZALES I, PARAMODIAZ M. LONG-TERM RESULTS OF RESTORATIVE ARTERIAL SURGERY IN OBSTRUCTIVE DISEASES OF THE ARTERIES. J Cardiovasc Surg (Torino). 1964 Nov-Dec;5:463-72. No abstract available. PMID 14242827
- [Background] Caraceni A, Cherny N, Fainsinger R, Kaasa S, Poulain P, Radbruch L, De Conno F. Pain measurement tools and methods in clinical research in palliative care: recommendations of an Expert Working Group of the European Association of Palliative Care. J Pain Symptom Manage. 2002 Mar;23(3):239-55. doi: 10.1016/s0885-3924(01)00409-2. PMID 11888722
- [Background] Frampton CL, Hughes-Webb P. The measurement of pain. Clin Oncol (R Coll Radiol). 2011 Aug;23(6):381-6. doi: 10.1016/j.clon.2011.04.008. Epub 2011 May 14. PMID 21571514
- [Background] Galer BS, Jensen MP. Development and preliminary validation of a pain measure specific to neuropathic pain: the Neuropathic Pain Scale. Neurology. 1997 Feb;48(2):332-8. doi: 10.1212/wnl.48.2.332. PMID 9040716
- [Background] Bonezzi C, Nava A, Barbieri M, Bettaglio R, Demartini L, Miotti D, Paulin L. [Validazione della versione italiana del Brief Pain Inventory nei pazienti con dolore cronico]. Minerva Anestesiol. 2002 Jul-Aug;68(7-8):607-11. Italian. PMID 12244292
- [Background] Negri E, Bettaglio R, Demartini L, Allegri M, Barbieri M, Miotti D, Paulin L, Buonocore M, Bonezzi C. [Validation of the Italian version of the "Neuropathic Pain Scale" and its clinical applications]. Minerva Anestesiol. 2002 Mar;68(3):95-104. Italian. PMID 11981518
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Charlson M, Szatrowski TP, Peterson J, Gold J. Validation of a combined comorbidity index. J Clin Epidemiol. 1994 Nov;47(11):1245-51. doi: 10.1016/0895-4356(94)90129-5. PMID 7722560
- [Background] Benyamin R, Trescot AM, Datta S, Buenaventura R, Adlaka R, Sehgal N, Glaser SE, Vallejo R. Opioid complications and side effects. Pain Physician. 2008 Mar;11(2 Suppl):S105-20. PMID 18443635
- [Derived] Venturini MA, Zappa S, Minelli C, Bonardelli S, Lamberti L, Bisighini L, Zangrandi M, Turin M, Rizzo F, Rizzolo A, Latronico N. MAGnesium-oral supplementation to reduce PAin in patients with severe PERipheral arterial occlusive disease: the MAG-PAPER randomised clinical trial protocol. BMJ Open. 2015 Dec 16;5(12):e009137. doi: 10.1136/bmjopen-2015-009137. PMID 26674497